Official Title of the Study: Nourish: A Pilot Study and Co-Design

NCT Number: NCT06398197

**Date of the Document**: June 27, 2024



# INFORMED CONSENT DOCUMENT Nourish Pilot Study: Cooking Classes

You are being asked to participate in a research study conducted by researchers at Case Western Reserve University. This consent form contains important information about this project and what to expect if you decide to participate. Please consider the information carefully. Feel free to ask questions before making your decision whether or not to participate. Your participation in this research is voluntary.

## **KEY INFORMATION FOR YOU TO CONSIDER:**

The **purpose of the research** study is to learn more about the best ways to teach cooking and food skills to adults, and the how cooking classes may help reduce one's stress and food waste, as well as improve their diet.

**Major study activities and expected duration of participation:** This study involves participating in cooking class over 8 weeks and completion of two rounds surveys. The maximum possible duration of this study is 20 weeks, but only 10 weeks of active participation.

**Why?** Other than possibly learning some new information and techniques, participating may not directly help you, but your participation may help researchers learn more about the best ways to teach cooking to adults and the how cooking classes may help reduce one's stress and food waste, as well as improve their diet.

Why Not? There is an unlikely possibility you may not like some of the questions or that they may make you uncomfortable. You can refuse to answer any of the questions, take a break, or stop your participation in this study at any time. There is a rare risk for a loss of confidentiality any time data is collected.

Please refer to the Detailed Consent for additional information.

#### **DETAILED CONSENT**

You were selected as a possible participant because you may be interested and able to attend in-person cooking classes within your community and are an adult at least 18 years of age. We hope to recruit 40 people to volunteer for this research. As part of this study, you will be randomized (similar to the flipping of a coin) to one of two study groups. One group will participate in the Nourish cooking class first and the second group will participate in the Nourish cooking class after the first group completes the class. You will be told which group you have been randomized to.

#### **First Survey Meeting:**

Regardless of which group you are in, you will participate in the first survey meeting. At this visit you will sign the consent form and complete surveys to better understand your access to food, food behaviors, and stress in your daily life.

You will also be asked to complete a series of two 24-hour dietary recalls (via phone calls) lasting approximately 30 minutes each and asked to weigh and log your food waste for one week.

Version 04/2021

During the first survey meeting, you will be asked to share your phone number and be given a kitchen food scale and waste log. You will return the log on the first day of the cooking class. Additionally, we will give you an overview of to expect at each Nourish class. In addition to the items described above, we are encouraging you to sign up for an app called GroupMe to receive out-of-class information about Nourish. The duration of the baseline assessment meeting will be approximately 60 minutes, and you will be told if you have been randomized to the immediate cooking class or delayed cooking class.

At the end of this meeting, you will be told a date and time when you will begin the cooking class.

#### **Nourish Cooking Class:**

The cooking class consists of eight 90 minute Nourish cooking classes. These cooking classes will take place in the teaching kitchen at Dave's Market (Midtown) or CornUcopia. Each class will involve brief instructional video clips, hands-on cooking and tasting experiences. You will work individually and as part of small groups during the instructional sessions. At the end of each class, you will receive a grocery bundle and a kitchen gadget to help you apply what you learned in class. After each Nourish Cooking Class, we will also ask you to complete a brief online, anonymous survey to provide feedback on each lesson, which will take approximately 10 minutes or less.

We will also ask you to post photos of what you made with your groceries to GroupMe. You will earn raffle tickets for each time you post to the GroupMe and attend a class. A raffle drawing for a pressure cooker will be done at the second survey meeting for the immediate cooking class group and at the final Nourish class for the delayed cooking class group.

The delayed intervention group will commence the Nourish intervention after the post-intervention assessment period is complete (i.e. ~2 weeks after the 8<sup>th</sup> class of the first cohort).

#### **Second Survey Meeting:**

Regardless of which group you are in, you will participate in the second survey meeting at week 10, which will last about 35 minutes. Two weeks prior to this meeting, you will be asked to complete a series of two 24-hour dietary recalls (via phone calls) lasting approximately 30 minutes each and asked to weigh and log your food waste for one week. During the meeting, you will be asked to repeat the survey complete about your access to food, food behaviors, and stress in your daily life.

You will also be asked to return the food waste log at the second survey meeting.

## **Foreseeable Risks and Discomforts**

All procedures may involve some level of risk to you. We have listed below the foreseeable risks, but there may be some that are unforeseeable.

Any time information is collected, there is a potential risk for loss of confidentiality. There are no other known risks of harms or discomforts associated with this study beyond those encountered in normal daily life. Some of the activities we will ask you to complete might make you feel uncomfortable. You may refuse to answer any of the questions, take a break, or stop your participation in this study at any time. Possible risks and/or discomforts associated with the procedures described in this study include boredom, emotional distress, etc.

## **Anticipated Benefits**

The possible benefits you may experience from the procedures described in this study include learning about nutrition, food safety, cooking, and meal preparation, and possibly managing stress through these activities. *IRB Version* 02/2023

Your participation in this study may help researchers learn more about the best ways to teach cooking to adults and the how cooking classes may help reduce one's stress and food waste, as well as improve their diet.

## **Compensation**

There will be no costs to you for study participation.

You will not be provided compensation or reimbursement for travel expenses, time off work or child care.

You will receive the following compensation:

| Immediate Cooking Class Group: | | | | | Delayed Cooking Class Group: | | |
|---|---|---|---|---|---|---|---|
| | | | Total | | | | Total |
| When | What | Compensation | cash | When | What | Compensation | Cash |
| First | Food/stress | \$35 | \$35 | First | Food/stress | \$35 | \$35 |
| Survey | Survey | | | Survey | Survey | | |
| Meeting | Diet | \$20 for each of 2 diet | \$40 | Meeting | Diet | \$20 for each of 2 diet | \$40 |
| | Interviews | interview phone calls | | | Interviews | interview phone calls | |
| Week 1 | Food waste tracking | \$50 for tracking one week's worth of food | \$50 | Week 1 | Food waste tracking | \$50 for tracking one week's worth of food | \$50 |
| | S | waste | | | | waste | |
| Nourish | Cooking | 8 cooking classes: each | | Nourish | | | |
| Classes | classes and | providing the opportunity | | Classes | | | |
| | class | to eat the cooked meal, a | | | | | |
| Weeks | feedback | cooking/kitchen gadget | | Weeks | | | |
| 3-10 | surveys | (\$15 value each class), | | 3-10 | Wi | Il not participate | |
| | | and small grocery bundle | \$40 | | | | \$0 |
| | | (\$15 value each class). | | | | | |
| | | 8 brief class feedback | | | | | |
| | | surveys (\$5 each) | | | | | |
| Second | Food | \$35 | \$35 | Second | Food | \$35 | \$35 |
| Survey | Survey | | | Survey | Survey | | |
| Meeting | Diet | \$20 for each of 2 diet | \$40 | Meeting | Diet | \$20 for each of 2 diet | \$40 |
| | Interviews | interview phone calls | | | Interviews | interview phone calls | |
| Week | Food waste | \$50 for tracking one | \$50 | Week | Food waste | \$50 for tracking one | \$50 |
| 12 | tracking | week's worth of food | | 12 | tracking | week's worth of food | |
| | | waste | | | | waste | |
| Nourish | | | | Nourish | Cooking | 8 cooking classes: each | |
| Classes | | | | Classes | classes and | providing the | |
| | | | | | class | opportunity to eat the | |
| Weeks | | | | Weeks | feedback | cooked meal, a | |
| 13-20 | *** | | 40 | 13-20 | surveys | cooking/kitchen gadget | <b></b> |
| | W | ill not participate | \$0 | | | (\$15 value each class), | \$40 |
| | | | | | | and small grocery | |
| | | | | | | bundle (\$15 value each | |
| | | | | | | class). | |
| | | | | | 8 brief class feedback | | |
| C | | | | Cua | | surveys (\$5 each) | |
| Grand | | | 6200 | Grand | | | 6200 |
| Total<br>Cash | | | \$290 | Total<br>Cash | | | \$290 |
| Cash | | | | Casn | | | |

Also, every time you complete an at-home cooking challenge and post your own photo of it to the group chat, you will be entered into a drawing to receive a pressure cooker.

If you decide to withdraw from the study or are withdrawn by the research team, you will receive compensation for the surveys and classes that you have completed.

## Alternative(s) to Participation

Participation is voluntary and you can stop participating at any time. There is no alternative to participating, other than not participating.

#### **Voluntary Nature of the Study**

Your participation is voluntary. If you choose not to participate, it will not affect your current or future relations with the University. There is no penalty or loss of benefits for not participating or for discontinuing your participation.

You are free to withdraw from this study at any time. If you decide to withdraw from this study, you should notify the research team immediately. The research team may also end your participation in this study if you do not follow instructions, miss scheduled visits, or if your safety or welfare are at risk.

If you elect to withdraw or are withdrawn from this research study, the researchers will discuss with you what will happen to your study data. The researchers will ask for your permission to retain and analyze the study data already collected. If the data collected are de-identified (anonymous) the researchers will not have the ability to remove your study data.

#### **Confidentiality**

Every effort will be made to keep your information confidential; however, this cannot be guaranteed. Research records will be kept in a secure location and access will be limited to the researchers, the University review board responsible for protecting human participants, regulatory agencies, and National Science Foundation. In any sort of report we might publish, we will not include any information that will make it possible to identify a participant.

However, you should understand that in cases where we suspect elder or child abuse or neglect or imminent harm to self or others, we will take the necessary action in an effort to prevent such harm or injury, including reporting to authorities.

**All** information that identifies you will be removed from the study data.

#### Data Retention

The researchers intend to keep the research data:

• For approximately 1 year after analysis of the information is completed

### **Contacts and Questions**

The researcher conducting this study is Dr. Melissa Prescott. You may ask any questions you have now. If you have any additional questions, concerns or complaints about the study, you may contact the researcher:

(216) 368-4699, melissa.prescott@case.edu

If you would like to talk to someone *other than the researchers* about questions or complaints regarding this study, research participant rights, research-related injuries, or other concerns, please contact: Case Western Reserve University Institutional Review Board

IRB Version 02/2023

10900 Euclid Ave. Cleveland, OH 44106-7230 (216) 368-4514 cwru-irb@case.edu

# **Statement of Consent**

Your signature below certifies the following:

- You are at least 18 years of age.
- You have read (or been read) the information provided above.
- You have received answers to all of your questions and have been told who to call if you have any more questions.
- You have freely decided to participate in this research.
- You understand that you are not giving up any of your legal rights.

| You will be given a copy of this form for your records. | |
|---------------------------------------------------------|-------|
| Printed Name of Participant | |
| Signature of Participant | Date: |
| Signature of Person Obtaining Consent | Date: |